CLINICAL TRIAL: NCT06123559
Title: Effects of Physical Exercise and Motor Activity on Depression and Anxiety in Post-Mastectomy Pain Syndrome
Brief Title: Physical Exercise, Motor Activity and Depression in Post-mastectomy Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Other Study IDs: BCMADA
Record Dates: First submitted 2023-10-17; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain
Keywords: Chronic pain; post mastectomy; depression; anxiety; motor activity; haematological markers
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Pain is an unpleasant sensation common to all those who undergo surgery. Several studies indicate that 40-60% of patients experience the post-operative experience and can be caused by both internal and external stimuli. Chronic post mastectomy pain is a condition characterized by pain in the anterior chest, armpit, and/or upper arm, usually ipsilateral to surgery, which begins after mastectomy or quadrantectomy and persists for longer three months after surgery. It can become chronic in a broad spectrum of conditions. Psychosocial factors such as anxiety and catastrophizing are being revealed as crucial contributors to individual differences in pain processing and outcomes. Some researchers have reported the associations between the development of persistent pain catastrophizing and depression or psychological distress and reduced physical activity. Taken together, these symptoms may lead to disability and worsened quality of life. Due to its benefits, the American Cancer Society recommends to begin as soon as possible from the diagnosis of cancer, physical activity. Aim of this prospective observational study is to evaluate the effects of motor and/or sports activity on the intensity of chronic pain and in symptoms of depression and anxiety, caused by post-mastectomy chronic pain. of life of women underwent mastectomy.

DETAILED DESCRIPTION:
Chronic pain is one of the most frequent occurring after surgery. It leads to functional limitations and psychological disorders, with a negative impact on quality of life.

Chronic post-surgical pain (CPSP) was first defined as "pain that develops after surgical intervention and lasts at least 2 months; other causes of pain have to be excluded, in particular, pain from a condition existing before the surgery".

An updated definition of CPSP, or persistent post-surgical pain (PPSP), was later proposed by Werner and Kongsgaard in 2014. The proposed definition was "pain persisting at least three months after surgery, that was not present before surgery, or that had different characteristics or increased intensity from preoperative pain, localized to the surgical site or a referred area, and other possible causes of the pain were excluded (e.g., cancer recurrence, infection)".

Persistent post-mastectomy pain (PPMP) is a major individual and public health problem. The etiology of persistent pain after mastectomy is still unclear, although it is likely multifactorial and may be partially of neuropathic origin. While surgical factors, including more extensive surgery (total vs partial mastectomy), axillary lymph node dissection, and reconstruction, have been postulated to serve as important risk factors for chronic pain, many studies do not support this association. Adjuvant treatment, such as radiation, chemotherapy, and hormone therapy, has also been occasionally associated with persistent pain.It is estimated that 25-60% of patients who have undergone breast cancer removal surgery suffer from PMP syndrome and psychosocial factors such as anxiety, depression, sleep disturbance and catastrophizing have proven to be important contributors to the development of persistent pain . A link between pain and depression is well known, it is suggested that 30%-45% of patients affected by chronic pain, experience depression. Several studies have suggested a bidirectional relationship between depression and pain, suggesting that depression is a positive predictor of the development of chronic pain and chronic pain can increases the risk of developing depression. Moreover depression is considered a moderator of the relationship between pain severity and physical functioning . It is known that depressive disorders overlap with anxiety disorders, anxiety symptoms are included in the diagnostic criteria for major depressive disorder in the diagnostic and statistical manual of mental disorders 5th edition (DSM-5). Results obtained from from case control studies suggest that inflammation could be involved in generalized anxiety disorder, indicating that inflammation could increase subsequent to the development of an anxiety disorder.

The aim of this study was to evaluate the effects of physical activity on the intensity and interference of chronic pain in daily activities and the effect on depression and anxiety in patient underwent mastectomy.

Study population: women underwent unilateral or bilateral mastectomy due to resection of stage II and III breast cancer not followed by breast reconstruction aged 18 years or older who have not received chemotherapy or radiation. Pain assessment: Pain assessment is a multidimensional process, which must take into account all the components of suffering, both physically, psychologically and socially. The assessment of pain and motor activity of each participant in the study will be carried out 3 and 6 months after surgery. Pain will be assessed by administration of Numerical Rating Scale (NRS) questionnaire. For the evaluation of depression, was used the Beck's Depression Inventory (BDI) and for the anxiety evaluation, will be administered the Generalized Anxiety Disorders-7 (GAD-7). All the evaluation will be performed 3 and 6 months after surgery.

The IPAQ (International Physical Activity Questionnaire) questionnaire measures the type and amount of physical activity that is normally done. The questions refer to the activity carried out in the last 7 days. It will be administered at 3 and 6 months after surgery.The expected duration of the study can be considered to be approximately 12 months. At the same time-points (12 and 24 weeks after surgery) biomarkers of pain, inflammation and correlated to anxiety and depression will be measured together with routine blood parameters. Specifically, the following biomarkers will be evaluated: IL-17, IL-1beta, brain-derived neutrophic factor (BDNF), cortisol and adrenocorticotropic hormone (ACTH).

ELIGIBILITY:
Inclusion Criteria: over the age of 18 with a diagnosis of previous Stages I-III breast cancer

Exclusion Criteria:

* medical history of other types of cancer;
* disease related to the immune system (e.g. multiple sclerosis, HIV, lupus);
* recent symptoms of illness (cough, fever);
* no antinflammatory or antidepressive or anxiolitic drugs assumption during the first six months after surgery
* waiting breast reconstruction;
* not chemotherapy or radiation during the first six months after surgery:

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women underwent unilateral or bilateral mastectomy due to resection of stage II and III breast cancer.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Effects of motor and/or sports activity on the intensity of chronic pain in women underwent mastectomy. | Evaluation performed three and six months after surgery
  Pain intensity self-measured using the Numerical Rating Scale (NRS). NRS is a 0-11 point-scale where the end points are the extremes of no pain (point 0) and worst pain as bad as it could be (point 10).
Effects of motor and/or sports activity on depression in women underwent mastectomy suffering by chronic pain. | Evaluation performed three and six months after surgery
  Depression will be evaluated with Beck's Depression Inventory (BDI) questionnaire. BDI consists of twenty-one questions about how the subject has been feeling in the last week. Each question has at least four possible answer choices; a value of 0 to 3 is assigned for each answer and then the total score determines the severity of depression as follow: 0-9: indicates normal or minimal depression; 10-18: indicates mild depression; 19-29: indicates moderate depression; 30-63: indicates severe depression.
Effects of motor and/or sports activity on anxiety in women underwent mastectomy suffering by chronic pain. | Evaluation performed three and six months after surgery
  Anxiety will be evaluated with Generalized Anxiety Disorders-7 (GAD-7) questionnaire. Each item asks the individual to rate the severity of his or her symptoms over the past two weeks. A score of 0, 1, 2, and 3 is assigned to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21 described as follow: 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety.

SECONDARY OUTCOMES:
Evaluation of biomarker associated to pain intensity, depression and anxiety | Evaluation performed three and six months after surgery]
  Biomarkers correlated to pain intensity, depression and anxiety, were evaluated in serum. Analysis was performed in blood aliquot withdrawn during the routine analysis. The following biomarkers were considered: IL-17 (pg/mL), IL-1beta (pg/mL), ACTH (pg/mL) and BDNF (pg/mL). All the measures were performed by ELISA according to the manufacturer protocol.
Evaluation of serum cortisol | Evaluation performed three and six months after surgery
  Serum cortisol (ng/mL) was evaluated by ELISA analysis, according to the manufaturer protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Gioacchino Calapai, Messina, Italy

REFERENCES:
- [Background] Zhang JM, An J. Cytokines, inflammation, and pain. Int Anesthesiol Clin. 2007 Spring;45(2):27-37. doi: 10.1097/AIA.0b013e318034194e. PMID 17426506
- [Background] Calapai M, Esposito E, Puzzo L, Vecchio DA, Blandino R, Bova G, Quattrone D, Mannucci C, Ammendolia I, Mondello C, Gangemi S, Calapai G, Cardia L. Post-Mastectomy Pain: An Updated Overview on Risk Factors, Predictors, and Markers. Life (Basel). 2021 Sep 29;11(10):1026. doi: 10.3390/life11101026. PMID 34685397
- [Background] Ambrose KR, Golightly YM. Physical exercise as non-pharmacological treatment of chronic pain: Why and when. Best Pract Res Clin Rheumatol. 2015 Feb;29(1):120-30. doi: 10.1016/j.berh.2015.04.022. Epub 2015 May 23. PMID 26267006
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Schreiber KL, Martel MO, Shnol H, Shaffer JR, Greco C, Viray N, Taylor LN, McLaughlin M, Brufsky A, Ahrendt G, Bovbjerg D, Edwards RR, Belfer I. Persistent pain in postmastectomy patients: comparison of psychophysical, medical, surgical, and psychosocial characteristics between patients with and without pain. Pain. 2013 May;154(5):660-668. doi: 10.1016/j.pain.2012.11.015. Epub 2012 Dec 5. PMID 23290256
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Hodes GE, Kana V, Menard C, Merad M, Russo SJ. Neuroimmune mechanisms of depression. Nat Neurosci. 2015 Oct;18(10):1386-93. doi: 10.1038/nn.4113. Epub 2015 Sep 25. PMID 26404713
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Alderman BL, Olson RL, Brush CJ, Shors TJ. MAP training: combining meditation and aerobic exercise reduces depression and rumination while enhancing synchronized brain activity. Transl Psychiatry. 2016 Feb 2;6(2):e726. doi: 10.1038/tp.2015.225. PMID 26836414
- [Background] Archer T, Josefsson T, Lindwall M. Effects of physical exercise on depressive symptoms and biomarkers in depression. CNS Neurol Disord Drug Targets. 2014;13(10):1640-53. doi: 10.2174/1871527313666141130203245. PMID 25470398
- [Background] Maes M, Abe Y, Sirichokchatchawan W, Suwimonteerabutr J, Sangkomkamhangd U, Almulla AF, Satthapisit S. The Cytokine, Chemokine, and Growth Factor Network of Prenatal Depression. Brain Sci. 2023 Apr 26;13(5):727. doi: 10.3390/brainsci13050727. PMID 37239199